CLINICAL TRIAL: NCT06678139
Title: The Effect of a Physiotherapy on Lower Extremity Function and Gait in Children with Isolated Gastrocnemius Muscle Tightness
Brief Title: The Effect of Physiotherapy on Lower Extremity Function and Gait in Children with Isolated Gastrocnemius Muscle Tightness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant Professor, Bezmialem Vakif University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12.10.2024-168536
Record Dates: First submitted 2024-11-04; First posted 2024-11-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-11

CONDITIONS: Lower Extremity Biomechanics; Gastrocnemius Tightness; Pes Planovalgus
Keywords: Isolated gastrocnemius muscle tightness; physiotherapy; lower extremity function; gait
MeSH Terms: conditions — Clubfoot | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Exercise group
  Interventions: Other: physiotherapy

INTERVENTIONS:
Other: physiotherapy — Bilateral gastrosoleus stretching, iliopsoas and hamstring stretching (if a shortness is detected), foot intrinsic and extrinsic muscle strengthening, lower extremity muscle strengthening and parkour walking training will be performed. Therapeutic exercises will be performed once a week for 12 weeks under the supervision of a physiotherapist. Parents will be asked to follow a 12-week home exercise program at home during the five days. The home exercise program will include the exercises performed in the pediatric physiotherapy and research laboratory. Parents will be instructed to perform each exercise twice a day at home. Children will be given a weekly exercise diary to increase adherence to the exercise program.

SUMMARY:
Since the gastrocnemius muscle crosses both joints, the joint kinematics of the ankle are affected by knee flexion. According to the Kendall & McCreary assessment of normal joint motion angles, the generally accepted normal range of motion for ankle dorsiflexion is 20° when the knee joint is in extension and can approach 30° when the knee joint is flexed due to relaxation of the gastrocnemius. In the mid-stance phase of gait, it is observed that the ankle joint allows 8-10° dorsi flexion movement.

In this study, a minimum 13° increase in dorsiflexion with knee flexion compared to dorsiflexion with knee extension will be considered as isolated gastrocnemius muscle tightness. Isolated gastrocnemius muscle tightness has been associated with many biomechanical changes such as pes planus, talar equinus, hindfoot pronation and symptoms such as plantar fasciitis, leg pain, metatarsalgia, achilles tendinopathy by compensatory effects on the lower extremity and foot during gait. The association of increased hindfoot pronation with isolated gastrocnemius tightness has been shown in many studies. Regardless of the etiology of pronation of the hindfoot, there will be adaptive isolated gastrocnemius tightness with talar plantar flexion. Isolated gastrocnemius tightness, which causes plantar flexion in the ankle joint and pronation in the subtalar joint, also prevents the distribution of the load to the base of the foot within normal limits during weight bearing. However, no study investigating the effect of physiotherapy program on function and gait has been encountered. The aim of this study was to investigate the effect of a physiotherapy program on lower extremity function and gait in children with isolated gastrocnemius muscle tightness.

ELIGIBILITY:
Inclusion Criteria:

* Presence of bilateral pes planovalgus due to the isolated gastrocneius tightness
* Being the ages between 4-10 years old
* Having body mass index between within normal limits

Exclusion Criteria:

* Presence of high femoral anteversion (Craig test > 30 degrees) and/or internal tibial torsion and/or metatursus adductus
* Having of leg length discrepancy
* Accompanying any neurological, rheumatologic, musculoskeletal, metabolic and connective tissue disease
* Presence of pain associated with the vertebral column and lower extremities
* Presence of any lower extremity and/or vertebral column deformity or history of surgery
* Cognitive, mental, serious psychiatric illness
* Participation in any exercise program and/or sportive activity in the last six months

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-03-22 (Actual); Study Completion 2025-03-22 (Actual)

PRIMARY OUTCOMES:
Gait analyses with Kinovea ® software | Baseline and immediately after the physiotherapy program
  The following assessments will be carried out before starting the exercise program. Then the children will be positioned at the beginning of the prepared 5-meter walking path with their underwear on. First, they will be asked to take trial walks and then they will be asked to walk 5 times on this path at their normal walking pace. Video recordings will be taken from frontal (antero-posterior) and sagittal (lateral) planes with a camera placed on a tripod. The same assessments and video recordings will be repeated at the end of the 12-week physiotherapy program. Observational gait analysis will be performed by scoring with the Edinburg Observational Gait Scoring using the frame-by-frame tracking feature of the video. Video recordings of the children obtained from 3 different angles (anterior-posterior-lateral) will be monitored and scored in slow motion with Kinovea ® software
Edinburgh Observational Gait Score | Baseline and immediately after the physiotherapy program
  The Edinburgh Observational Gait Score is an easy-to-use, reliable visual scoring system. In 2003, Read et al. developed this scoring system by identifying the key points of pathologic gait in CP. It has 17 parameters evaluating gait in sagittal, coronal and transverse planes, selected in association with computerized gait analysis. It allows the evaluation of archived gait videos for trunk, pelvis, hip, knee, ankle and foot according to the phases of gait.
Lower Extremity Function Scale | Baseline and immediately after the physiotherapy program
  It is a test completed by the parents to assess health-related quality of life. It includes some activities that require the use of the foot and leg in daily life. The degree of difficulty of the child with isolated gastrocnemius muscle tightness to perform these activities is scored between 0 (not difficult) and 4 (unable). As the test score gets closer to 0 (zero), the functional level of the child increases.

SECONDARY OUTCOMES:
Foot Posture Index (FPI-6) | Baseline and immediately after the physiotherapy program
  It is a practical method that provides information about the alignment disorders of the foot and allows evaluation in multiple plans. FPI-6 is a scoring system in the range of -12 and +12 obtained by scoring the data in the range of +2 and -2 for 6 separate analyzes. The evaluation will be performed in the position in which the children feel comfortable, with their arms at their sides, in a standing posture while looking straight ahead. Each analysis will be scored on a 5-point scale (+2, +1, 0, -1, -2) with positive values indicating pronation and negative values indicating supination.
Navicular Drop Test | Baseline and immediately after the physiotherapy program
  The navicular drop test is a test used clinically to determine the presence and degree of pes planus. In this test, the navicular tubercle is first palpated and marked and the distance between the navicular tubercle and the floor is measured while the person is in a sitting position and the feet are only in contact with the floor (without weight on the feet). The distance between the navicular tubercle and the floor is then measured again with the person standing up and putting equal weight on the feet. Measurements will be made bilaterally and recorded in millimeters (mm). In the navicular drop test, the difference between weighted and unweighted measurements between 5-9 mm is considered normal (neutral), 10 mm or more is considered pronation, and 4 mm or less is considered supination.
Sit to Stand Test | Baseline and immediately after the physiotherapy program
  The child will be asked to get up from a chair without armrests and sit back down again with his/her hips and knees flexed at 90° and feet in full contact with the floor. The number of sit-ups within 30 seconds will be recorded with a stopwatch.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tuncer D, Eren Zengin F, Senaran H, Uzer G. The effect of a 12-week physiotherapy program on lower extremity function and gait in children with isolated gastrocnemius tightness. Physiother Theory Pract. 2025 Dec;41(12):2605-2616. doi: 10.1080/09593985.2025.2542415. Epub 2025 Aug 6. PMID 40767345